CLINICAL TRIAL: NCT01125969
Title: A Randomized Trial of Incentives and Peer Mentors to Improve Diabetic Outcomes
Brief Title: A Trial of Incentives and Peer Mentors to Improve Diabetic Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 10022605
Record Dates: First submitted 2010-04-13; First posted 2010-05-19 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; glucose; peer mentor; incentives; behavioral economics; cost-effectiveness
MeSH Terms: conditions — Diabetes Mellitus | interventions — Fertility; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator)
  Interventions: Behavioral: Education
- Incentive (Experimental)
  Interventions: Behavioral: Incentives; Behavioral: Education
- Peer Mentoring (Experimental)
  Interventions: Behavioral: Education; Behavioral: Peer mentoring
- Incentives and Peer Mentoring (Experimental)
  Interventions: Behavioral: Incentives; Behavioral: Education; Behavioral: Peer mentoring

INTERVENTIONS:
Behavioral: Incentives — Incentives will be offered for checking blood glucose each morning and for control of blood glucose (between 80-140 mg/dL).
  Arms: Incentive; Incentives and Peer Mentoring
Behavioral: Education — Standard brochure about improving blood sugar control plus warnings about dangers of persistently high sugars and hypoglycemia
Behavioral: Peer mentoring — Participant is assigned a peer mentor who is matched on gender, race and age and who achieved good glucose control after previously having poor glucose control.
  Arms: Incentives and Peer Mentoring; Peer Mentoring

SUMMARY:
In recent years, social networks have garnered attention in both academic journals and the lay press because of strong associations demonstrated in retrospective studies between social networks and incidence of major health problems such as obesity and smoking. Financial incentives have also been demonstrated to improve health behaviors in obesity, smoking, and medication adherence. We propose to conduct a randomized controlled trial among a predominantly African American population with persistently poor diabetes mellitus (DM) control to examine whether two novel interventions, lottery based financial incentives and telephone based one-on-one peer mentoring (the 'buddy system'), can significantly ameliorate disparities in poor DM control.

The intervention is based on epidemiologic evidence, randomized controlled trials, and pilot studies demonstrating: 1) Lottery based financial incentives are a powerful motivator of behavior change; 2) One-on-one peer mentoring is a flexible, cost-efficient means of increasing DM specific social support and may be particularly salient in minority communities; and 3) Matching patients with poorly controlled DM with a similar individual from their community who has gained control of their DM draws on existing community assets in creating an inherently culturally competent intervention. DM patients with poor DM control will be randomized to 1 of 4 arms: usual care; telephone based one-on-one peer mentoring; lottery based financial incentives; and peer mentoring plus financial incentives.

The Specific Aims are to test: 1) The effectiveness of telephone based one-on-one peer mentoring in improving glycemic control relative to usual care; 2) The effectiveness of lottery based financial incentives in improving glycemic control relative to usual care; 3) The effectiveness of combining peer mentoring and financial incentives relative to control; and 4) The relative cost effectiveness of all four approaches. In exploratory analyses, we will examine whether African American patients enrolled in intervention arms have greater improvement in glycemic control than white patients, whether intervention group patients experience greater improvements in blood pressure (BP) and lipid control, and whether peer mentors experience improvements in their own health. We will pair mentors with mentees based on race, gender, age, and disease severity. The active intervention will be run for a 6-month time period, with participants followed for an additional 6 months to determine if effects persist post intervention.

The proposed interventions address multiple barriers to effective disease management common among patients with DM. If effective, these interventions could provide important models for improving glycemic control in general and, in particular, for addressing racial disparities in DM outcomes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with diabetes mellitus
* 30 to 70 years old
* persistently poor glucose control, defined as having the last two HbA1c values > 8%, with at least one measure within 3 months of enrollment
* receiving treatment for diabetes mellitus at one of five University of Pennsylvania outpatient clinics

Exclusion Criteria:

* does not speak English
* unable to provide informed consent

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | Baseline, 6 months
  HbA1c is a measure of the percent of glycosylated hemoglobin in the blood stream. It is an excellent biomarker reflecting glucose control for the preceding 2-3 months and thus provides a reliable and unbiased marker of patient adherence. The primary outcome will be a change in HbA1c from baseline to the 6-month follow-up visit.

SECONDARY OUTCOMES:
Cost-effectiveness of change in Hemoglobin A1c | 6 months
  A "within-trial" analysis will be conducted that adopts the perspective of an insurer and directly compares costs and change in HbA1c using data measured in the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Judith A. Long, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States